CLINICAL TRIAL: NCT06793007
Title: Anatomical Variants of Intrahepatic Bile Ducts and Cystic Duct in Magnetic Resonance Cholangiopancreatography: A Retrospective Cross-Sectional Study in a Tertiary Hospital in Kathmandu.
Brief Title: Variants Of Intrahepatic Biliary Radicals in Nepali Population
Acronym: IHBR
Status: Completed | Type: Observational
Sponsor: Grande International Hospital, Nepal (Other)
Responsible Party: Principal Investigator, PRAJWAL DAHAL, Principal Investigator, Grande International Hospital, Nepal
Other Study IDs: 12/2024
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Liver Dysfunction
MeSH Terms: conditions — Liver Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic resonance imaging cholangiopancreatography

SUMMARY:
Biliary anatomical variations are commonly observed during diagnostic imaging and, if overlooked, can lead to considerable risks during surgical, endoscopic, or other interventional procedures. In Nepal, where advanced imaging techniques such as MRCP are becoming more accessible, it is crucial to understand the prevalence and types of these variants within the local population. This understanding aids in enhancing pre-surgical planning, minimizing surgical complications, and improving diagnostic precision. By analyzing retrospective data from a private hospital, this study aims to provide important insights into regional anatomical variations, supporting improved clinical outcomes.

DETAILED DESCRIPTION:
Anatomy of the biliary tree is intricate, with numerous intrahepatic and extrahepatic variations and cystic duct variations that are crucial to recognize to avoid complications in surgical or interventional procedures (1,2). Detailed anatomical knowledge is essential as bile duct surgeries, liver resections, and transplants become increasingly sophisticated (1). Magnetic Resonance Cholangiopancreatography (MRCP) is a preferred non-invasive imaging technique that safely and accurately maps both the bile and cystic duct anatomy without radiation exposure, ideal for patients with contrast allergies (2). Intrahepatic bile ducts follow the portal veins, with the right hepatic duct draining segments 5, 6, 7, and 8 and the left hepatic duct draining segments 2, 3, and 4. The right and left hepatic ducts merge at the hilum to form the CHD. With standard branching patterns occurring in roughly 50-60% of cases, knowledge of these frequent variants is critical for safe and effective surgical planning (4).

The classification of the right hepatic duct (RHD) by Huang et al. (2) includes five types: Type A1 (classic, RPD and RAD form RHD), Type A2 (trifurcation, all ducts converge), Type A3 (RPD drains into LHD), Type A4 (RAD drains into CHD), and Type A5 (absent RHD). Karakas et al. similarly classify the RHD into five types, mirroring Huang's types with slight variations in naming conventions. The left hepatic duct (LHD) classification by Cho A et al. (2) consists of four types: Type I (classic, LHD drains into RHD), Type II (accessory duct from the left lateral segment), Type III (segmental ducts join RHD or CHD separately), and Type IV (no unified LHD formation). These classifications are essential for understanding anatomical variations relevant to hepatobiliary surgeries and MRCP imaging.

Typically, the cystic duct is 2-4 cm long and 1-5 mm in diameter, joining the gallbladder neck to the common hepatic duct (CHD) to form the common bile duct (CBD), usually entering the CHD from the right lateral side (4). Variations in the cystic duct's insertion, length, and course-including low or high insertion points, parallel courses with the CHD, spiral orientations, and occasionally absent ducts-are documented and clinically significant (4).

There are few studies of similar kind done in Nepali population. Sharma et al(1)studied the prevalences of different variants of right hepatic duct as per classification of choi et al in 90 patients. In their study, 47.8% of patients were classified as having Type 1/normal intrahepatic bile duct (IHBD) variations (n=43). Type 2 was observed in 20% of the cases (n=18), while Type 3A accounted for 3.3% (n=3) and Type 3B for 5.6%. Type 5A was present in 5 patients (n=5), and Type 5B in 7.8% (n=7), with Type 6 seen in 3.3% (n=3) and Type 7 in 6.7% (n=6). No cases of Type 3C or Type 4 variations were identified. Among the Type 1 patients, 67.44% (n=29) were female, while the remainder were male. Sarawagi R(2) et al conducted a study similar to ours and obtained the prevalences of variants of right hepatic duct as per classification by Huang et al. The right posterior sectoral duct (RPSD) draining into the left hepatic duct (LHD) was the most common variant, observed in 27.6% of subjects. A trifurcation pattern was noted in 9.3% of cases, while 4% of subjects had the RPSD draining into the common hepatic duct (CHD) and 0.8% into the cystic duct. Other variants were seen in 2.6% of subjects, and an accessory duct was present in 4.9% of cases. The most frequent branching pattern of the LHD was a common trunk formed by the segment 2 and 3 ducts joining the segment 4 duct, seen in 67.8% of subjects. In 23.2% of subjects, the segment 2 duct united with the common trunk of segments 3 and 4, while 3.4% had all three segments (2, 3, and 4) merging to form the LHD. Other less common branching patterns were observed in 4.9% of subjects.K.C et al(3) studied about variants of cystic duct in Nepali population in 252 patients. The most frequently observed type was the right lateral insertion, found in 120 patients (47.62%), while the remaining patients exhibited other anatomical variants. The posterior insertion was the second most common variant, seen in 36 patients (14.29%), followed by high insertion in 25 patients (9.92%). The right posterior sectoral hepatic duct draining into the cystic duct was the least common variant. Sarawagi et al(4) also studied about variants of cystic duct in MRCP in Indian population. Normal lateral insertion of the cystic duct (CD) at the middle third of the common hepatic duct was found in 51% of cases. Medial insertion was seen in 16% (4% low medial), while low insertion occurred in 9%. A parallel course of the CD was present in 7.5%, high insertion in 6%, and a short CD in 1%. In one case, the CD drained into the right hepatic duct, and another case exhibited congenital cystic dilation consistent with a type IV choledochal cyst.

The four studies collectively highlight the diversity and prevalence of anatomical variations in the biliary system across different populations. Variations in the right hepatic duct were common, with normal intrahepatic bile duct patterns (Type 1) being the most prevalent, seen in 47.8% of cases in Sharma et al.'s study, while Sarawagi et al. noted that the right posterior sectoral duct (RPSD) draining into the left hepatic duct was the most frequent variant (27.6%). Trifurcation patterns and accessory ducts were also observed but were less common. Regarding cystic duct variants, both K.C. et al. and Sarawagi et al. found that the lateral insertion into the common hepatic duct was the most prevalent pattern, seen in 47.62% and 51% of cases, respectively. Other common variations included posterior and high insertions of the cystic duct, while rare cases such as RPSD draining into the cystic duct and congenital cystic dilation were also documented. These findings underscore the significance of understanding these variations for clinical and surgical applications.

ELIGIBILITY:
Inclusion Criteria:

* All high quality, diagnostically adequate MRCP scans of patients age > 18 years done in our department for various indications an no previous hepatobiliary surgery (except cholecystectomy)are included in the study

Exclusion Criteria:

* Diagnostically inadequate, unclear MRCP scans were excluded from the study. Also, scans of patient < 18 years, patients with hepatobiliary surgery and pathology distorting normal anatomy were also excluded. Scans with biliary obstruction were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of all gender and age 18 and above
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of different variants on intrahepatic biliary radicals | 6 months
  Prevalence of different variants on intrahepatic biliary radicals in Nepali population

CONTACTS AND LOCATIONS:
Locations (1):
- Tokha Road, Dhapasi, Kathmandu, Bagmati, Nepal

REFERENCES:
- [Background] 1. Paudel S, Joshi BR, Chand RB. Evaluation of Intrahepatic Bile Duct Variations in Magnetic Resonance Cholangiopancreatography. Nepal J Radiol. 2020 Dec 1;10(1):27-33.
- [Background] Sarawagi R, Sundar S, Raghuvanshi S, Gupta SK, Jayaraman G. Common and Uncommon Anatomical Variants of Intrahepatic Bile Ducts in Magnetic Resonance Cholangiopancreatography and its Clinical Implication. Pol J Radiol. 2016 May 26;81:250-5. doi: 10.12659/PJR.895827. eCollection 2016. PMID 27298653
- [Background] 3. Kc S, Banjade UR, Ghimire P. Anatomical variations of the cystic duct assessed by magnetic resonance cholangiopancreatography (MRCP): a cross-sectional study at tertiary center of Nepal. J Patan Acad Health Sci. 2024 Jun 14;11(1):15-20.
- [Background] Sarawagi R, Sundar S, Gupta SK, Raghuwanshi S. Anatomical Variations of Cystic Ducts in Magnetic Resonance Cholangiopancreatography and Clinical Implications. Radiol Res Pract. 2016;2016:3021484. doi: 10.1155/2016/3021484. Epub 2016 May 25. PMID 27313891